CLINICAL TRIAL: NCT04374136
Title: A Phase 3, Multicenter, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of AL001 in Individuals at Risk for or With Frontotemporal Dementia Due to Heterozygous Mutations in the Progranulin Gene
Brief Title: A Phase 3 Study to Evaluate Efficacy and Safety of AL001 in Frontotemporal Dementia (INFRONT-3)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial did not meet the clinical co-primary endpoint of slowing FTD-GRN progression, as measured by the Clinical Dementia Rating® plus National Alzheimer's Coordinating Center Frontotemporal Lobar Degeneration Sum of Boxes (CDR® plus NACC FTLD-SB)
Sponsor: Alector Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL001-3
Record Dates: First submitted 2020-04-23; First posted 2020-05-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Frontotemporal Dementia
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AL001 (Experimental): AL001 every 4 weeks
  Interventions: Drug: AL001
- Placebo (Placebo Comparator): Placebo every 4 weeks
  Interventions: Drug: Placebo
- Open label - AL001 (Experimental): AL001 every 4 weeks
  Interventions: Drug: Open label - AL001

INTERVENTIONS:
Drug: AL001 — Administered via intravenous (IV) infusion
  Arms: AL001
Drug: Placebo — Administered via intravenous (IV) infusion
  Arms: Placebo
Drug: Open label - AL001 — Administered via intravenous (IV) infusion
  Arms: Open label - AL001

SUMMARY:
A phase 3 double blind, placebo controlled study evaluating the efficacy and safety of AL001 in participants at risk for or with frontotemporal dementia due to heterozygous mutations in the progranulin gene.

DETAILED DESCRIPTION:
This is a phase 3 double blind, placebo controlled study evaluating the efficacy and safety of AL001 administered intravenously in participants at risk for or with frontotemporal dementia due to heterozygous mutations in the progranulin gene. Study completion marks the end of the open label extension period following the 96-week blinded portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a progranulin gene mutation and at risk of developing FTD symptoms as evidenced by a biomarker, or persons with a progranulin gene mutation and diagnosed with FTD.
* If symptomatic, one or more of the criteria for the diagnosis of possible behavioral variant FTD, or a diagnosis of Primary Progressive Aphasia.
* Study partner who consents to study participation and who cares for/visits the participant daily for at least 5 hours per week.
* Written informed consent must be obtained and documented (from the participant or, where jurisdictions allow it, from their legal decision maker).

Exclusion Criteria:

* Dementia due to a condition other than FTD including, but not limited to, Alzheimer's disease, Parkinson's disease, dementia with Lewy bodies, Huntington disease, or vascular dementia.
* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins.
* Current uncontrolled hypertension, diabetes mellitus or thyroid disease. Clinically significant heart disease, liver disease or kidney disease. History or evidence of clinically significant brain disease other than FTD.
* Females who are pregnant or breastfeeding, or planning to conceive within the study period.
* Any experimental vaccine or gene therapy.
* History of cancer within the last 5 years.
* Current use of anticoagulant medications (e.g., coumadin, heparinoids, apixaban).
* Residence in a skilled nursing facility, convalescent home, or long term care facility at screening; or requires continuous nursing care.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of AL001 as measured by the CDR® plus NACC FTLD-SB | Through study completion, on average up to 96 weeks
  The Clinical Dementia Rating Dementia Staging Instrument PLUS National Alzheimer's Disease Coordinating Center frontotemporal lobar degeneration Behavior & Language Domains Sum of Boxes (CDR® plus NACC FTLD-SB) is administered by a healthcare professional and based on individual ratings of the eight domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, personal care, language and behavior. Impairment is scored on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2 and severe = 3. The 8 individual domain ratings, or "box scores", were added together to give the CDR® plus NACC FTLD-SB which ranges from 0-24. Higher score indicates severe impairment.

SECONDARY OUTCOMES:
Change in Clinical Global Impression-Severity (CGI-S) Score | Baseline to 96 weeks
  The CGI-S is used by a clinician to rate the severity of a participant's disease relative to the clinician's past experience with patients who have the same disease using an ordinal scale ranging from 1=normal, not at all ill; 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill patients. Higher scores indicate worsening.
Change in Clinical Global Impression-Improvement (CGI-I) Score | Baseline to 96 weeks
  The CGI-I is used by a clinician to rate how much a participant's disease has improved or worsened relative to baseline using an ordinal scale ranging from 1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; and 7=very much worse. Higher scores indicate worsening.
Change in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Score | Baseline to 96 weeks
  RBANS is 20 to 25 minute battery developed for cognitive assessment, detection, and characterization of dementia. RBANS includes 12 subtests that measure following 5 indices: (1)Attention Index, composed of Digit Span and Coding; (2)Language Index, consisting of Picture Naming and Semantic Fluency subtests; (3)Visuospatial/Construction Index, made up of Figure Copy and Line Orientation subtests; (4)Immediate Memory Index, composed of List Learning and Story Memory subtests, and (5)Delayed Memory Index, consisting of List Recall, List Recognition, Story Recall, and Figure Recall subtests. Completion of RBANS yields 5 index scores based on participant performance on various subtests, as well as a composite Total Index score for battery. Total index scores range from 40 to 160, and are normalized to a mean of 100 and standard deviation (SD) of 15. Higher scores indicate less impairment.
Pharmacodynamic Biomarkers | Baseline to 96 weeks
  Change in magnetic resonance imaging and blood-based biomarkers and optional CSF biomarkers (neurofilament light chain and progranulin)
Evaluation of safety and tolerability of AL001: Incidence of adverse events | Baseline to 96 weeks
  Incidence of adverse events

OTHER OUTCOMES:
Optional Open-Label Extension | 96 weeks
  Assess the long-term safety and tolerability of AL001 in participants who have completed 96 week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, Principal Investigator
Locations (44):
- United States (14):
  - Dignity Health, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas Alzheimer's Disease Center, Fairway, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Mayo Comprehensive Cancer Center - PPDS, Rochester, Minnesota
  - Irving Institute for Clinical and Translational Research, New York, New York
  - University Of Cincinnati Gardner Neuroscience institute, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Institute for Academic Medicine, Houston, Texas
- Fundación Para La Lucha Contra Las Enfermedades Neurológicas de La Infancia, Buenos Aires, Argentina
- Australia (2):
  - Box Hill Hospital, Box Hill
  - The Queen Elizabeth Hospital, Woodville
- UZ Leuven, Leuven, Vlaams Brabant, Belgium
- Canada (2):
  - The University of Western Ontario, London
  - Sunnybrook Research Institute - University of Toronto, Toronto
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHRU Lille, Lille
  - Groupe Hospitalier Pitié Salpétrière, Paris
- Germany (2):
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - Eginitio University General Hospital of Athens - 1st University Neurology Clinic, Athens, Attica
  - University General Hospital of Alexandroupolis - Department of Neurology, Alexandroupoli, Evros
- Italy (6):
  - Nuovo Ospedale Civile S. Agostino-Estense di Baggiovara, Baggiovara
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia
  - IRCCS - Centro S. Giovanni di Dio Fatebenefratelli, Brescia
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta, Milan
  - PIA Fondazione Panico, Tricase
- Erasmus MC, Rotterdam, Netherlands
- Portugal (4):
  - Centro Hospitalar E Universitário de Coimbra EPE, Coimbra
  - Centro Hospitalar de Lisboa Norte, EPE - Hospital de Santa Maria, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian
- Karolinska Universitetssjukhuset Huddinge - PPDS, Huddinge, Sweden
- Felix Platter Spital, Basel, Switzerland
- Istanbul University Medical Faculty, Istanbul, Fatih, Turkey (Türkiye)
- University College London, London, United Kingdom